CLINICAL TRIAL: NCT03709628
Title: An Open-label, Multicenter, Pharmacokinetic Study of a FimH Blocker, EB8018, in Crohn's Disease Patients
Brief Title: A Study of a FimH Blocker, EB8018, in Crohn's Disease Patients
Acronym: EBFIM117
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enterome (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Enterome
Record Dates: First submitted 2018-04-11; First posted 2018-10-17 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with active Crohn's disease (Experimental): EB8018: 3000 mg for the single dose in Part 1 (2 sentinel patients) and 1500 mg BID for multiple dose administration over 13 days in Parts 1 and 2 (2 sentinel patients and 6 remaining patients), oral.
  Interventions: Drug: EB8018 (First-in-class FimH blocker)

INTERVENTIONS:
Drug: EB8018 (First-in-class FimH blocker) — Drug: EB8018 EB8018 is an orally administered, first-in-class, FimH blocker
  • In Part 1, a single oral dose of EB8018 3000 mg will be administered to the 2 sentinel patients in the morning on Day 1. In the multi-dose treatment period (part 1 and 2), multiple oral doses of EB8018 1500 mg will be administered to 2 + 6 patients BID (in the morning and evening) on Days 1 through 13.
  Other Names: EB8018

SUMMARY:
Enterome small molecule drug EB8018 is a first-in-class FimH blocker to be studied in Crohn's disease patients. The proposed indication for EB8018, as an add-on therapy, will be the treatment of adult patients suffering from Crohn's disease.

DETAILED DESCRIPTION:
This open-label, multicenter study will enroll 8 evaluable patients with active Crohn's disease and will consist of 2 parts. Part 1 will include 2 sentinel patients with a single dosing period followed by a 13-day multiple dosing period. Part 2 will include the 6 remaining patients with multiple dosing only. This Phase 1b study will investigate the PK, safety, preliminary effects of the gut microbiome, and inflammatory biomarkers of EB8018 following 13 days of consecutive BID oral dosing in patients with Crohn's disease.

Part 1 of this study will demonstrate a single oral dose of EB8018 that is safe and tolerable in patients with Crohn's disease and Part 2 of this study will characterize the PK profile when administered as multiple oral doses.

ELIGIBILITY:
Selection Criteria:

* Male and female patients of nonchildbearing potential ≥18 years of age at screening and Day -1
* Active Crohn's disease based on an elevated calprotectin at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Cmax | Day1, Day13
  Maximum observed plasma concentration
Tmax | Day1
  Time to maximum observed plasma concentration
AUC0-24 | Day1; Day13
  Area under the plasma concentration time curve from time 0 to 24 hours
T1/2 | Day1; Day13
  Terminal elimination half-life

SECONDARY OUTCOMES:
AE | Up to Day22
  Adverse events
RR | Up to Day22
  Inter-Beat intervalle (sec)
QRS complex | Up to Day22
  intervalle (sec)
QT | Up to Day22
  duration (sec)
PR | Up to Day22
  intervalle (sec)
HR | Up to Day22
  Heart rate (bpm)
BP | Up to Day22
  Blood pressure (mmHg)
RR | Up to Day22
  Respiratory rate (breaths per minute)
Temp | Up to Day22
  Temperature (C°)

OTHER OUTCOMES:
Gut Microbiome | Up to Day22
  Overall gene richness and relative abundance of Bacteroidetes, Enterobacteriaceae, and Firmicutes from sequencing of stool samples.
Inflammatory Biomarkers | Up to Day22
  C-reactive protein
Inflammatory Biomarkers | Up to Day22
  Fecal calprotectin
CDAI score | Up to Day22
  CDAI calculation will be dependent on the parameters recorded in the subjects' diary and the parameters assessed at clinic visit by the investigator.

CONTACTS AND LOCATIONS:
Locations (5):
- Medical University Vienna, Vienna, Austria
- France (2):
  - Hôpital Claude Huriez, Lille
  - Hôpital de l'Archet 2, Nice
- Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel, Germany
- Istituto Clinico Humanitas, Rozzano, Italy